CLINICAL TRIAL: NCT03415386
Title: A Multi-center Study on the Optimized Antithrombotic Therapy of Acute Myocardial Infarction With Left Ventricular Mural Thrombus.
Brief Title: Optimized Antithrombotic Therapy of Acute Myocardial Infarction With Left Ventricular Mural Thrombus
Acronym: OATH-AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: OATH-AMI
Record Dates: First submitted 2018-01-11; First posted 2018-01-30 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Acute Myocardial Infarction; Left Ventricular Thrombus
MeSH Terms: interventions — Anticoagulants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- aspirin100mg qd+clopidogrel75mg qd+warfarin (INR1.8-2.2) (Experimental)
  Interventions: Drug: Combination of antiplatelet drugs and anticoagulants for at least one month
- aspirin100mg qd+clopidogrel75mg qd+dabigatran110mg bid (Experimental)
  Interventions: Drug: Combination of antiplatelet drugs and anticoagulants for at least one month
- aspirin100mg qd+ticagrelor60mg bid+warfarin(INR1.8-2.2) (Experimental)
  Interventions: Drug: Combination of antiplatelet drugs and anticoagulants for at least one month
- aspirin100mg qd+ticagrelor60mg bid+dabigatran110mg bid (Experimental)
  Interventions: Drug: Combination of antiplatelet drugs and anticoagulants for at least one month

INTERVENTIONS:
Drug: Combination of antiplatelet drugs and anticoagulants for at least one month — Combination of antiplatelet drugs and anticoagulants for at least one month, such as aspirin100mg qd+clopidogrel75mg qd+warfarin (INR1.8-2.2), aspirin100mg qd+clopidogrel75mg qd+dabigatran110mg bid, aspirin100mg qd+ticagrelor60mg bid+warfarin (INR1.8-2.2), and aspirin100mg qd+ticagrelor60mg bid+dabigatran110mg bid. Transthoracic two-dimensional echocardiography will be done at the 1-month, 3-month and 6-month follow-ups to evaluate the left ventricular mural thrombus and determinate whether the antithrombotic therapy regimen could be regulated to double antiplatelet or anticoagulant+clopidogrel75mg qd/ticagrelor60mg bid.

SUMMARY:
A multi-center study will be done to explore the optimal regimen of antithrombotic therapy for acute myocardial infarction with left ventricular mural thrombus. The investigators will evaluate the different combinations of antiplatelet drugs and anticoagulants for at least one month, such as aspirin 100mg qd+clopidogrel 75mg qd+warfarin (INR1.8-2.2), aspirin 100mg qd+clopidogrel 75mg qd+dabigatran 110mg bid, aspirin 100mg qd+ticagrelor 60mg bid+warfarin (INR1.8-2.2), and aspirin 100mg qd+ticagrelor 60mg bid+dabigatran 110mg bid. Transthoracic two-dimensional echocardiography will be done at the 1-month, 3-month and 6-month follow-ups to evaluate the left ventricular mural thrombus and determinate whether the antithrombotic therapy regimen could be regulated to double antiplatelet or anticoagulant+clopidogrel 75mg qd/ticagrelor 60mg bid. Then the investigators will complete the 12-month follow-up to evaluate the efficacy and safety of the optimal antithrombotic therapy regimen for acute myocardial infarction with left ventricular mural thrombus.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction with left ventricular mural thrombus

Exclusion Criteria:

* BARC bleedings ≥ 2
* atrial fibrillation
* acute stroke or other systemic circulation embolism

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mural thrombus-1 | 1-month
  Number of Participants Without left ventricular mural thrombus as Assessed by echocardiograph at 1-month.
Left ventricular mural thrombus-3 | 3-month
  Number of Participants Without left ventricular mural thrombus as Assessed by echocardiograph at 3-month.
Left ventricular mural thrombus-6 | 6-month
  Number of Participants Without left ventricular mural thrombus as Assessed by echocardiograph at 6-month.

SECONDARY OUTCOMES:
Death | 12 months
Recurrent myocardial infarction | 12 months
Stroke or other systemic circulation embolism | 12 months
Stent restenosis | 12 months
Target vessel revascularization | 12 months
Major cardio-cerebral vascular events | 12 months
  Composite of any events from outcome 2 to 6

OTHER OUTCOMES:
Major bleeding | 12 months
  Bleeding Academic Research Consortium (BARC) bleedings ≥ 2
Minor bleeding | 12 months
  BARC bleedings < 2

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Reeder GS, Lengyel M, Tajik AJ, Seward JB, Smith HC, Danielson GK. Mural thrombus in left ventricular aneurysm: incidence, role of angiography, and relation between anticoagulation and embolization. Mayo Clin Proc. 1981 Feb;56(2):77-81. PMID 7464234
- [Background] Turpie AG, Robinson JG, Doyle DJ, Mulji AS, Mishkel GJ, Sealey BJ, Cairns JA, Skingley L, Hirsh J, Gent M. Comparison of high-dose with low-dose subcutaneous heparin to prevent left ventricular mural thrombosis in patients with acute transmural anterior myocardial infarction. N Engl J Med. 1989 Feb 9;320(6):352-7. doi: 10.1056/NEJM198902093200604. PMID 2643772
- [Background] Keeley EC, Hillis LD. Left ventricular mural thrombus after acute myocardial infarction. Clin Cardiol. 1996 Feb;19(2):83-6. doi: 10.1002/clc.4960190203. PMID 8821415